CLINICAL TRIAL: NCT03314181
Title: A Phase 1/2, Multicenter, Dose-Escalation and Expansion Study of Combination Therapy With Venetoclax, Daratumumab and Dexamethasone (With and Without Bortezomib) in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Combination Therapy With Venetoclax, Daratumumab and Dexamethasone (With and Without Bortezomib) in Participants With Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-654; 2017-002099-26 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2017-10-11; First posted 2017-10-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: t(11,14) positive relapsed/refractory (R/R) multiple myeloma; Non-refractory Relapsed Multiple Myeloma; Non-refractory Refractory Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma; Multiple Myeloma; Cancer; Venetoclax; Venclexta
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — Dexamethasone; daratumumab; venetoclax; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Arm A, Part 1a: VenDd Dose Escalation (Experimental): Venetoclax (Ven) various doses administered orally, once daily (QD) in combination with daratumumab (D) (1800 mg subcutaneous injection (preferred) or 16 mg/kg intravenous [IV]) administered in accordance with prescribing information and dexamethasone (d) (oral or IV) 40 mg weekly (or 20 mg weekly, if necessary, as described in the protocol).
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Venetoclax
- Arm B, Part 1b: VenDd Dose Expansion (Experimental): Venetoclax at a dose determined by the dose-escalation phase, administered orally QD in combination with daratumumab (1800 mg subcutaneous injection (preferred) or 16 mg/kg IV) administered in accordance with prescribing information and dexamethasone (oral or IV) 40 mg weekly (or 20 mg weekly, if necessary, as described in the protocol).
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Venetoclax
- Arm D, Part 2a: VenDVd Dose Escalation (Experimental): Venetoclax at various doses administered orally QD in combination with daratumumab (1800 mg subcutaneous injection (preferred) or 16 mg/kg IV) administered in accordance with prescribing information, bortezomib (1.3 mg/m2 subcutaneous injection [preferred] or IV) Cycles 1-8, Days 1, 4, 8 and 11), and dexamethasone (oral or IV) 20 mg Cycles 1 - 3, Days 1, 2, 4, 5, 8, 9, 11,12 and 15; 20 mg Cycles 4-8, Days 1,2,4,5,8,9,11 and 12; 40 mg weekly (or 20 mg weekly, if necessary as described in the protocol) Cycle 9+.
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Venetoclax; Drug: Bortezomib
- Arm E, Part 2b: VenDVd Dose Expansion (Experimental): Venetoclax at dose determined by the dose-escalation phase, administered orally QD in combination with daratumumab (1800 mg subcutaneous injection (preferred) or 16 mg/kg IV) administered in accordance with prescribing information, bortezomib (1.3 mg/m2 subcutaneous injection) Cycles 1-8, Days 1, 4, 8 and 11, and dexamethasone (oral or IV) 20 mg Cycles 1 - 3, Days 1, 2, 4, 5, 8, 9, 11,12 and 15; 20 mg Cycles 4-8, Days 1,2,4,5,8,9,11 and 12; 40 mg weekly (or 20 mg weekly, if necessary as described in the protocol) Cycle 9+.
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Venetoclax; Drug: Bortezomib
- Arm F: VenDd Dose Expansion (Experimental): Venetoclax at a pre-determined dose, administered orally QD in combination with daratumumab (1800 mg subcutaneous injection (preferred) or 16 mg/kg IV) administered in accordance with prescribing information and dexamethasone (oral or IV) 40 mg weekly (or 20 mg weekly, if necessary, as described in the protocol).
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Venetoclax
- Arm G: VenDd Dose Expansion (Experimental): Venetoclax at a pre-determined dose, administered orally QD in combination with daratumumab (1800 mg subcutaneous injection (preferred) or 16 mg/kg IV) administered in accordance with prescribing information and dexamethasone (oral or IV) 40 mg weekly (or 20 mg weekly, if necessary, as described in the protocol).
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Venetoclax
- Arm H: DVd Dose (Active Comparator): Daratumumab (1800 mg subcutaneous injection (preferred) or 16 mg/kg IV) administered in accordance with prescribing information, bortezomib (1.3 mg/m2 subcutaneous injection) Cycles 1-8: Days 1, 4, 8 and 11, and dexamethasone (oral or IV) 20 mg on Cycles 1 - 3: Days 1, 2, 4, 5, 8, 9, 11,12 and 15; 40 mg weekly (or 20 mg weekly, if necessary as described in the protocol) on Cycles 4-8: Days 1,2,4,5,8,9,11 and 12; 20 mg monthly for Cycles 9+: Day 1
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Bortezomib

INTERVENTIONS:
Drug: Dexamethasone — Infusion; Intravenous (IV), or Tablet; Oral
Drug: Daratumumab — Injection; Subcutaneous (preferred), Infusion; Intravenous (IV)
Drug: Venetoclax — Tablet; Oral
  Other Names: ABT-199; Venclexta
  Arms: Arm A, Part 1a: VenDd Dose Escalation; Arm B, Part 1b: VenDd Dose Expansion; Arm D, Part 2a: VenDVd Dose Escalation; Arm E, Part 2b: VenDVd Dose Expansion; Arm F: VenDd Dose Expansion; Arm G: VenDd Dose Expansion
Drug: Bortezomib — Injection; Subcutaneous (preferred), Infusion; Intravenous (IV)
  Arms: Arm D, Part 2a: VenDVd Dose Escalation; Arm E, Part 2b: VenDVd Dose Expansion; Arm H: DVd Dose

SUMMARY:
This is a study of venetoclax, daratumumab, and dexamethasone with and without bortezomib combination therapy to evaluate safety, tolerability, and efficacy of these combinations in participants with relapsed or refractory multiple myeloma. The study will consist of 3 distinct parts: Part 1 includes participants with t(11;14) positive relapsed/refractory (R/R) multiple myeloma who will receive venetoclax in combination with daratumumab and dexamethasone (VenDd); Part 2 includes participants with R/R multiple myeloma who will receive venetoclax in combination with daratumumab, bortezomib, and dexamethasone (VenDVd); Part 3 includes participants with t(11;14) positive R/R multiple myeloma who will receive venetoclax in combination with daratumumab and dexamethasone (VenDd) or daratumumab, bortezomib, and dexamethasone (DVd).

Part 1 and Part 2 are non-randomized and will be initiated with a dose-escalation phase in which increasing doses of venetoclax will be given with fixed doses of daratumumab and dexamethasone (Part 1a) or with fixed doses of daratumumab, bortezomib, and dexamethasone (Part 2a). Each dose escalation phase will be followed by a single-arm, open-label expansion phase. Part 3 will include a randomized, open-label expansion phase with participants receiving venetoclax in combination with daratumumab and dexamethasone (VenDd) or daratumumab, bortezomib, and dexamethasone (DVd).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status <= 2.
* Participant has relapsed or refractory multiple myeloma with documented evidence of progression that occurred during or after the participant's last treatment regimen based on investigator's determination of International Myeloma Working Group (IMWG) criteria.
* Measurable disease confirmed by central lab at Screening, defined by at least 1 of the following: Serum M-protein >= 1.0 g/dL (>= 10 g/L), OR Urine M-protein >= 200 mg/24 hours, OR Serum free light chain (FLC) >= 10 mg/dL, provided serum FLC ratio is abnormal in participants who do not have measurable disease by Serum Protein Electrophoresis (SPEP) or Urine Protein Electrophoresis (UPEP) criteria.
* Participant has received previous multiple myeloma treatment as defined in the protocol.
* Bone marrow aspirate samples have been collected.
* To qualify for Part 1 and 3, the participant must be t(11;14) positive as determined by an analytically validated Fluorescent In Situ Hybridization (FISH) assay per central laboratory testing.
* Participants must have adequate hematologic, renal and hepatic function.

Exclusion Criteria:

* Previous treatment with venetoclax or other B-Cell Lymphoma 2 (BCL-2) inhibitor
* For participants in Parts 1 and 2: Previous treatment with daratumumab or other anti-CD38 therapy. For participants in Part 3: Prior daratumumab or other anti-CD38 antibody therapy exposure that meets ANY of the following criteria:

  * Failure to achieve at least a PR to most recent therapy with daratumumab or other anti-CD38 therapy.
  * Daratumumab or other anti-CD38 antibody therapy was discontinued due to toxicity.
  * Relapse within 60 days of intensive treatment (at least every other week) of daratumumab or other anti-CD38 antibody therapy.
  * Prior treatment with daratumumab or other anti-CD38 antibody within 6 months prior to first dose of study drug.
* For participants in Part 2 and 3:

  * Participant is refractory to any proteasome inhibitor, defined as progression on or within 60 days of the last dose of a proteasome inhibitor-containing regimen.
  * Participant has had prior treatment with proteasome inhibitor within 60 days prior to first dose of study drug.
* Treatment with anti-myeloma chemotherapy, radiotherapy, biological, immunotherapy or an investigational therapy, including targeted small molecule agents within 2 weeks or 5 half-lives (whichever is longer and/or applicable) before first dose.
* Treatment with anti-myeloma monoclonal antibodies within 6 weeks prior to first dose.
* Recent corticosteroid therapy at a cumulative dose equivalent to >= 140 mg of prednisone, cumulative dose equivalent to >= 40 mg of dexamethasone, or a single dose equivalent to >= 40 mg of dexamethasone within 2 weeks prior the first dose of study drug.
* Known central nervous system involvement of multiple myeloma.
* Significant history of medical conditions as listed in the protocol.
* History of other active malignancies including myelodysplatic syndromes (MDS) within the past 3 years with the exceptions of:

  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin.
  * Prostate cancer Gleason grade 6 or lower AND with stable Prostate Specific Antigen (PSA) levels off treatment
  * Previous malignancy with no evidence of disease confirmed and surgically resected (or treated with other modalities) with curative intent and unlikely to impact survival during the duration of the study.
* Known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* Has a hypersensitivity or allergy to any of the components of study therapy, excipient or boron.
* Known allergies, hypersensitivities, or intolerance to monoclonal antibodies or human proteins, or their excipients, or known sensitivity to mammalian-derived products (see daratumumab prescribing information).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2031-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 3.5 years after the last participant is enrolled
  ORR is defined as the percentage of participants with documented partial response (PR) or better based on International Myeloma Working Group (IMWG) criteria.
Very Good Partial Response or Better Response Rate (VGPR) | Up to approximately 3.5 years after the last participant is enrolled
  VGPR or better response rate is defined as the proportion of participants with documented VGPR or better (sCR, CR. or VGPR) based on IMWG criteria.
Complete Response (CR) or Better Rate | Up to approximately 3.5 years after the last participant is enrolled
  CR or better response is defined as the percentage of participants with documented response of CR or better (stringent complete response [sCR] or CR) based on IMWG criteria.
Time to Response (TTR) | Up to approximately 3.5 years after the last participant is enrolled
  TTR is defined as the number of days from the date of treatment start (for subjects enrolled prior to randomization start) or randomization (for randomized subjects) to the date of first documented response of PR or better.
Duration of Response (DOR) | Up to approximately 3.5 years after the last participant is enrolled
  DOR is defined as the number of days from the participant's date of first documented response (PR or better) to the date of first documented disease progression or death due to multiple myeloma, whichever occurs first.
Time to Progression (TTP) | Up to approximately 3.5 years after the last participant is enrolled
  TTP is defined as the number of days from the date of treatment start (for subjects enrolled prior to randomization start) or randomization (for randomized subjects) to the date of first documented PD or death due to MM, whichever occurs first.
Progression-Free Survival (PFS) | Up to approximately 3.5 years after the last participant is enrolled
  PFS is defined as the number of days from the date of treatment start (for subjects enrolled prior to randomization start) or randomization (for randomized subjects) to the date of the first documented PD or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 3.5 years after the last participant is enrolled
  OS is defined as the number of days from the date of treatment start (for subjects enrolled prior to randomization start) or randomization (for randomized subjects) to the date of death.

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) | Up to 12 months after confirmation of Complete Response (CR) or Stringent Complete Response (sCR)
  MRD negativity in bone marrow aspirates is defined at 10^-5 threshold as assessed by next generation sequencing (NGS) in participants at the time of suspected CR/sCR, and at 6 and 12 months post confirmation of CR/sCR for participants who maintained this response.
Cmax of Venetoclax | Up to approximately 1 year
  Maximum observed plasma concentration (Cmax) of venetoclax
Tmax of Venetoclax | Up to approximately 1 year
  Time to Cmax (Tmax) of Venetoclax
AUC0-24 of Venetoclax | Up to approximately 1 year
  Area under the plasma concentration-time curve (AUC) over the dose interval (AUC0-24) of venetoclax.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (40):
- United States (14):
  - Univ of Colorado Cancer Center /ID# 167331, Aurora, Colorado
  - Moffitt Cancer Center /ID# 169614, Tampa, Florida
  - Winship Cancer Institute of Emory University /ID# 165427, Atlanta, Georgia
  - The University of Chicago Medical Center /ID# 165429, Chicago, Illinois
  - Beth Israel Deaconess Medical Center /ID# 210904, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 166886, Boston, Massachusetts
  - Hackensack Univ Med Ctr /ID# 225111, Hackensack, New Jersey
  - Duplicate_Roswell Park Comprehensive Cancer Center /ID# 169615, Buffalo, New York
  - Weill Cornell Medicine/NYP /ID# 167605, New York, New York
  - Atrium Health Carolinas Medical Center /ID# 164948, Charlotte, North Carolina
  - Duke Cancer Center /ID# 165104, Durham, North Carolina
  - Duplicate_Wake Forest Baptist Health /ID# 224447, Winston-Salem, North Carolina
  - Oregon Health and Science University /ID# 166822, Portland, Oregon
  - University of Washington /ID# 164884, Seattle, Washington
- Australia (7):
  - The Kinghorn Cancer Centre /ID# 165431, Darlinghurst, New South Wales
  - St George Hospital /ID# 171063, Kogarah, New South Wales
  - Duplicate_Royal Adelaide Hospital /ID# 171060, Adelaide, South Australia
  - Eastern Health /ID# 165850, Box Hill, Victoria
  - St Vincent's Hospital Melbourne /ID# 165853, Fitzroy Melbourne, Victoria
  - Peter MacCallum Cancer Ctr /ID# 164742, Melbourne, Victoria
  - Duplicate_Royal Perth Hospital /ID# 224895, Perth, Western Australia
- Canada (3):
  - Arthur J. E. Child Comprehensive Cancer Centre /ID# 167822, Calgary, Alberta
  - Cross Cancer Institute /ID# 203114, Edmonton, Alberta
  - Disc_Royal Victoria Hospital / McGill University Health Centre /ID# 167824, Montreal, Quebec
- Denmark (4):
  - Rigshospitalet /ID# 164420, Copenhagen Ø, Capital Region
  - Duplicate_Aarhus University Hospital /ID# 164509, Aarhus N, Central Jutland
  - Odense University Hospital /ID# 164417, Odense, Region Syddanmark
  - Sygehus Lillebalt, Vejle /ID# 164418, Vejle, Region Syddanmark
- France (6):
  - CHU Limoges - Dupuytren 1 /ID# 224759, Limoges, Franche-Comte
  - CHRU Tours - Hopital Bretonneau /ID# 164795, Tours, Indre-et-Loire
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 164767, Nantes, Pays de la Loire Region
  - Institut Gustave Roussy /ID# 164807, Villejuif, Val-de-Marne
  - CHU Poitiers - La miletrie /ID# 164806, Poitiers, Vienne
  - Duplicate_AP-HP - Hopital Saint-Louis /ID# 224758, Paris
- Germany (2):
  - Universitaetsklinikum Freiburg /ID# 166036, Freiburg im Breisgau, Baden-Wurttemberg
  - University Hospital Cologne /ID# 166037, Cologne, North Rhine-Westphalia
- Japan (4):
  - Nagoya City University Hospital /ID# 225273, Nagoya, Aichi-ken
  - Kameda General Hospital /ID# 225246, Kamogawa-shi, Chiba
  - Duplicate_Matsuyama Red Cross Hospital /ID# 225196, Matsuyama, Ehime
  - Gifu Municipal Hospital /ID# 240381, Gifu, Gifu

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Bahlis NJ, Baz R, Harrison SJ, Quach H, Ho SJ, Vangsted AJ, Plesner T, Moreau P, Gibbs SD, Coppola S, Yang X, Al Masud A, Ross JA, Bueno O, Kaufman JL. Phase I Study of Venetoclax Plus Daratumumab and Dexamethasone, With or Without Bortezomib, in Patients With Relapsed or Refractory Multiple Myeloma With and Without t(11;14). J Clin Oncol. 2021 Nov 10;39(32):3602-3612. doi: 10.1200/JCO.21.00443. Epub 2021 Aug 13. PMID 34388020
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — http://www.rxabbvie.com